CLINICAL TRIAL: NCT00351949
Title: IMP321 Phase 1 Study in Advanced or Metastatic Renal Cell Carcinoma Patients (P003)
Brief Title: IMP321 Phase 1 Trial in Metastatic Renal Cell Carcinoma (MRCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Collaborators: Umanis (Industry)
Responsible Party: F. Triebel, Chief Medical Officer, Immutep S.A.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P003; Umanis-CRO0306
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Stage IV Renal Cell Carcinoma
Keywords: Advanced or metastatic renal cell carcinoma; IMP321; Monotherapy; LAG-3; CD223
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — soluble LAG-3 protein, human

INTERVENTIONS:
Biological: IMP321 — subcutaneous injections of IMP321 every 14 days for three months (6 injections. Doses tested: 50, 250, 1,250, 6,250 or 30,000 µg
  Other Names: hLAG-3Ig; LAG-3

SUMMARY:
Single-center, open label, non-randomized, fixed dose-escalation, phase 1 study, performed in ambulatory and day-hospital setting

DETAILED DESCRIPTION:
This is a single-center, single-arm, open label, non-randomized, fixed dose-escalation, phase 1 study, performed in ambulatory and day-hospital setting. After a screening period, patients will enter a drug administration period, followed by a 'post-study' period.

Four IMP321 dose levels, 50 µg, 250 µg, 1.250 mg, 6.250 mg and 30 mg will be evaluated in successive cohorts of patients. At any given dose level 3 patients will be administered one subcutaneous dose every 2 weeks for a total of 12 weeks (6 injections in total), separated by 13-day administration-free intervals.

The next (higher) dose level will be dosed to 3 new patients if the previous dose level has been well tolerated. Investigator will decide whether the safety is acceptable by performing an evaluation after the third administration (at week 8) and if the next patients can be included.

The successive cohorts of patients are summarized as follows:

* Cohort A will correspond to a group of 3 patients receiving the 50 µg dose. If safety at this dose level is acceptable as evaluated a fortnight after the 6-week administration, the following cohort will be undertaken.
* Cohort B will correspond to a group of 3 patients receiving the 250 µg dose. If safety at this dose level is acceptable as evaluated a fortnight after the 6-week administration, the following cohort will be undertaken.
* Cohort C will correspond to a group of 3 patients receiving the 1,250 µg dose. If safety at this dose level is acceptable as evaluated a fortnight after the 6-week administration, the following cohort will be undertaken.
* Cohort D will correspond to a group of 3 patients receiving the 1,250 µg dose. If safety at this dose level is acceptable as evaluated a fortnight after the 6-week administration, the following cohort will be undertaken.
* Cohort E will correspond to a group of 3 patients receiving the 6,250 µg dose. The patients will receive their first administration one-by-one with a two-weeks interval. If safety at this dose level is acceptable as evaluated a fortnight after the 6-week administration for the last patient, the following cohort will be undertaken.
* Cohort F will correspond to a group of 3 patients receiving the 6,250 µg dose. If the tolerability of this dose level has been judged acceptable in cohort E, the three patients will receive their first IMP321 injection simultaneously.
* Cohort G will correspond to a group of 3 patients receiving the 30,000 µg dose. The patients will receive their first IMP321 administration one-by-one with a two-weeks interval (+/- 5 days). If safety at this dose level is acceptable as evaluated a fortnight after the 6-week administration for the last patient, the following cohort will be undertaken.
* Cohort H will correspond to a group of 3 patients receiving the 30,000 µg dose. If the tolerability of this dose level has been judged acceptable in cohort E, the three patients will receive their first IMP321 injection simultaneously.

Once the main period of study has been completed, namely two weeks after a cohort is completed, i.e. at week 14, all patients will undergo an ambulatory 'post-study' examination.

Patients of the Cohort B, C, E, F and G will participate in a pharmacokinetic (PK) study and all patients in a pharmacodynamic (PD) study involving additional blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic renal clear cell (MRCC) adenocarcinoma, histologically proven by biopsy of the primary tumor and/or a metastasis. Prior nephrectomy is not required. The patient will be included in the study only if an efficacious cancer treatment can not be proposed.
* Patient to whom the currently available anticancer treatments are contra-indicated.
* Male or female 18 years or above. NB: Women must be either post-menopausal, rendered surgically sterile or practicing a reliable method of contraception (hormonal, intrauterine device or barrier). Pregnant women are excluded from this study.
* ECOG performance status 0-1.
* Expected survival longer than three months.
* Total white cell count ≥ 3.109/L.
* Platelet count ≥ 100.109/L.
* Hemoglobin > 9 g/dL or > 5.58 mmol/L.
* Serum creatinine < 160 µmol/L.
* Total bilirubin < 20 mmol/L, except for familial cholemia (Gilbert's disease)
* Serum ASAT and ALAT < 3 times the upper limit of normal or < 5 times upper limit of normal if liver metastases are present.
* Able to give written informed consent and to comply with the protocol.

Exclusion Criteria:

* Pregnancy, lactation or lack of effective contraception in fertile women of childbearing potential.
* Serious intercurrent infection within the 30 days prior to first administration.
* Known clinically active autoimmune disease.
* Known B or C active hepatitis.
* Known HIV positivity.
* Life threatening illness unrelated to cancer.
* Known cerebral metastases.
* Previous malignancies within the last two years other than successfully treated squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated with cone biopsy.
* Previous history of major psychiatric disorder requiring hospitalization or any current psychiatric disorder that would impede the patient's ability to provide informed consent or to comply with the protocol.
* Corticosteroids unless used as substitutive therapy.
* Past history of severe allergic episodes and/or Quincke edema.
* Past or present history of any organic disorder likely to modify absorption, distribution or elimination of the study drug.
* Alcohol or substance abuse disorder.
* IL-2 therapy or any other investigational agent within 30 days of first administration.
* Chemotherapy or radiotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first administration of the study drug or lack of recovery from adverse events (to grade 1 or less toxicity according to CTCAE 3.0) due to agents administered more than 4 weeks earlier. Exception is made regarding the x-ray treatment for painful bone metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Evaluate clinical and laboratory safety and tolerability profiles | 3 months
Determine pharmacokinetic and pharmacodynamic parameters | 3 months

SECONDARY OUTCOMES:
Secondary: Objective response rate (OR) using RECIST criteria | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Escudier, M.D, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Result] Brignone C, Escudier B, Grygar C, Marcu M, Triebel F. A phase I pharmacokinetic and biological correlative study of IMP321, a novel MHC class II agonist, in patients with advanced renal cell carcinoma. Clin Cancer Res. 2009 Oct 1;15(19):6225-31. doi: 10.1158/1078-0432.CCR-09-0068. Epub 2009 Sep 15. PMID 19755389
- See also: Sponsor's website — http://www.immutep.com